CLINICAL TRIAL: NCT04876794
Title: Clinical Investigation on Safety, Feasibility and Usability of the ABLE Exoskeleton Device With Spinal Cord Injured Patients in a Hospital Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ABLE Human Motion S.L. (Industry)
Collaborators: Institut Guttmann (Other); Heidelberg University Hospital Spinal Cord Injury Center (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABLEexoSCIhospital; CIV-20-07-034264 (Registry Identifier: EUDAMED)
Record Dates: First submitted 2021-04-30; First posted 2021-05-06 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-07

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injury; Exoskeleton; Robotics; Gait; Rehabilitation; Lower-limb; Neurorehabilitation; Paraplegia; Walking; Assistive technology; Usability; Safety; Feasibility; Multicenter
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Participants with SCI will undergo a training programme with the ABLE Exoskeleton device three times a week for four to six weeks for a total of 12 sessions.
  Interventions: Device: ABLE Exoskeleton

INTERVENTIONS:
Device: ABLE Exoskeleton — Participants with SCI will undergo a training programme with the ABLE Exoskeleton device three times a week for four to six weeks for a total of 12 sessions.

SUMMARY:
The loss of the ability to walk and the associated restriction of mobility presents a major challenge to people with spinal cord injury in an everyday environment designed for pedestrians. Exoskeletal technology has the potential to help people with impaired leg function to regain ambulation and thus improve their independence. This technology is not completely new, but due to their high access price (~120k€/unit), high size and weight (~25 kg), and need for trained physiotherapist supervision, commercially available exoskeletons are only found in large hospitals and only in very few cases get into patients' homes.

The company ABLE Human Motion S.L. (Barcelona, Spain) has developed a novel exoskeleton to overcome these disadvantages, which is more compact, lighter (9 kg) and easier to use.

The primary objective of the study is to investigate the safety, feasibility and usability of the ABLE exoskeleton device in people with spinal cord injury during a four to six weeks gait training in clinical settings. Furthermore, potential effects of the training on walking, general health status, user satisfaction, and quality of life will be assessed.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the safety, feasibility, and usability of using the ABLE Exoskeleton for patients with SCI in a hospital setting during a 4-6 week training programme.

The secondary objectives are as follows:

* Assess the impact of ABLE Exoskeleton training on gait and function.
* Assess the effect on the perceived rate of exertion for patients using the ABLE Exoskeleton.
* Assess the level of user satisfaction from participants and therapists of the ABLE Exoskeleton.
* Assess the psychosocial impact of the ABLE Exoskeleton for participants

Patients who match inclusion and exclusion criteria and pass pre-study screening will be enrolled in the study. Following the screening, baseline assessments will be conducted without the device. Participants will undergo a training programme with the ABLE Exoskeleton three times a week for four weeks for a total of 12 sessions. Standardized clinical assessments with the device will be performed during the first and the last training sessions. During the training period, several safety and usability measurements will be taken. After the last training session, baseline assessments without the exoskeleton will be repeated during a post-study assessment. Four weeks after the final training session a follow-up assessment will be conducted with participants. At the end of the study, the participating therapists will be asked to fill out a satisfaction questionnaire.

This is the first study investigating the use of the ABLE Exoskeleton, therefore the primary hypothesis of this study is that the ABLE Exoskeleton is safe, feasible, and usable for the intended patient population with SCI in a hospital setting. The secondary hypothesis is that the device will have a positive impact on the perceived rate of exertion, mobility, and psychosocial health of the study participants with SCI.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years of age
* Traumatic and non-traumatic SCI
* Currently receiving treatment as an inpatient or outpatient at one of the investigational sites
* AIS A to AIS D with sufficient arm strength to support body weight on a walking frame
* Ability to give informed consent

Exclusion Criteria:

* WISCI II without exoskeleton of >16
* 5 or more risk factors for fragility as stated by Craven et al (29)
* History of lower limb fragility fractures in the last 2 years
* Deterioration > 3 points of the total International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) motor score within the last 4 weeks
* Spinal instability
* Modified Ashworth scale (MAS) > 3 in lower limbs
* Unable to tolerate 30 min standing without clinical symptoms of orthostatic hypotension
* Unable to perform a sit-to-stand transfer or stand in the device with assistance
* Psychological or cognitive issues that do not allow a participant to follow the study procedures
* Any neurological condition other than SCI
* Medically unstable
* Severe comorbidities including any condition that a physician considers to not be appropriate to complete participation in the study
* Ongoing skin issues
* Height, width, weight or other anatomical constraints (such as leg length differences) incompatible with the device
* Insufficient Range of Motion (ROM) for ABLE Exoskeleton device
* Known pregnancy or breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
Safety | Up to 10 weeks
  To assess safety, the number of Severe Adverse Events (SAE), Adverse Events (AE) and drop-outs due to the device will be assessed and reported.
Time and Level of Assistance (LoA) to don/doff the device | Up to 8 weeks
  Level of Assistance (LoA) and time taken to don/doff the device will be measured in every session. LoA will be measured using a 6 item scale, from Total assistance to Independence. Different assistance levels are defined taking into account the degree of participation of both the patient and the therapist on performing the activity.
  This outcome measure will be used to assess the device's usability.
Level of Assistance (LoA) to complete therapy activity tasks | Up to 8 weeks
  Four therapy activity tasks will be attempted every session by the participant. The therapist will record the LoA required to complete each task during the session. The tasks are the following: sit-to-stand, walk 10 meters, turn 180 degrees, and stand-to-sit.
  Different assistance levels are defined taking into account the degree of participation of both the patient and the therapist in performing the activity.
  This outcome measure will be used to assess the device's usability.

SECONDARY OUTCOMES:
BORG Scale | Up to 7 weeks
  Measurement of the percieved rate of exertion. The BORG scale measures the subjective level of intensity in physical work on a 15-grade scale.
6-Minute Walk Test (6 MWT) | Up to 7 weeks
  6 Minute Walk Test (6 MWT) measures the distance a person can walk in 6 minutes. There are different possibilities for performing this test. For this study, we will use a track of 50 meters, where patients walk back and forth.
10-Meter Walking Test (10 MWT) | Up to 7 weeks
  The 10MWT will be performed using the first 10 meters of the 6-minute walking test.
Timed up and go test (TUG) | Up to 7 weeks
  Timed Up and Go Test (TUG) measures the time it takes a person to get up from a chair, walk 3 meters, turn around and sit down again. It is a widely used test to assess balance and the risk of falls in different patient groups.
Walking Index for Spinal Cord Injury (WISCI II) | Up to 7 weeks
  WISCI II assesses the extent and nature of assistance for walking 10 meters in persons with SCI. Assistance is specified as different combinations of braces, walking aids and physical assistance. The WISCI II consists of 20 levels from unable to walk to the ability to walk 10 meters without any assistance.
Spinal Cord Independence Measure (SCIM III) | Up to 10 weeks
  SCIM III scale focuses on the ability to perform activities of daily living in persons with SCI. The SCIM III consists of three subscales: Self-Care, Respiratory and Sphincter Management, Mobility (room and toilet) and Mobility (indoors and outdoors, on even surface). A total score of 0 (totally dependent) to 100 (totally independent) points can be achieved.
Quebec User Evaluation of Satisfaction with assistive Technology (QUEST 2.0) | Up to 10 weeks
  Used to measure user satisfaction from participants and therapists. QUEST 2.0 is designed to measure the level of satisfaction and the value people attribute to assistive technologies.
Psychosocial Impact of Assistive Devices Scale (PIADS) | Up to 10 weeks
  The PIADS is a 26-item (7-point Likert-Scale), self-report questionnaire designed to assess the effects of an assistive device on functional independence, well-being, and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Rüdiger Rupp, PD Dr., Principal Investigator — University Hospital Heidelberg
Locations (2):
- Spinal Cord Injury Center | Heidelberg University Hospital, Heidelberg, Germany
- Institut Guttmann, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No